CLINICAL TRIAL: NCT04513808
Title: Total IntraVenous AnesthesIa and ReCurrence-free Survival AfTer EsOphageal CanceR SurgerY
Brief Title: Total Intravenous Anesthesia and Recurrence Free Survival
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VICTORY
Record Dates: First submitted 2020-05-12; First posted 2020-08-14 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Intervention Model Description: As usual with time-to-event outcomes, enrollment will be based on the number of outcome events, not the number of patients enrolled. We anticipate that about 1614 patients will be required to generate 579 recurrences and/or deaths, but this is only a rough estimate since follow-up duration is a function of when patients are enrolled, not just their number.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol-based total intravenous anesthesia (Active Comparator): Propofol-based total intravenous anesthesia. A target-controlled infusion will be set to 2-4 µg/ml plasma concentrations, and varied as clinical necessary.
  Interventions: Drug: Propofol-based total intravenous anesthesia
- Sevoflurane intravenous anesthesia (Active Comparator): Anesthesia will be maintained with sevoflurane, typically at an end-tidal concentration of 0.6-1.0 MAC, but adjusted as clinically necessary
  Interventions: Drug: Sevoflurane intravenous anesthesia

INTERVENTIONS:
Drug: Propofol-based total intravenous anesthesia — Propofol-based total intravenous anesthesia, titrated to clinical need.
  Other Names: Propofol
  Arms: Propofol-based total intravenous anesthesia
Drug: Sevoflurane intravenous anesthesia — Sevoflurane intravenous anesthesia, titrated to clinical need.
  Other Names: Sevoflurane
  Arms: Sevoflurane intravenous anesthesia

SUMMARY:
The investigators propose to compare recurrence-free survival in patients having potentially curative (Stages 1-3) surgery for esophageal cancer who will be randomly assigned to propofol-based total intravenous anesthesia or sevoflurane-based balanced general anesthesia.

DETAILED DESCRIPTION:
The investigators will test the primary hypothesis that recurrence-free survival after esophageal cancer surgery is longer in patients randomized to propofol-based total intravenous anesthesia than to volatile sevoflurane anesthesia.

The investigators will test the secondary hypotheses that propofol-based total intravenous anesthesia: 1) speeds discharge from the ICU; 2) speeds discharge from the hospital; and, 3) improves the quality of recovery, as assessed by QoR-15 on postoperative day 2.

ELIGIBILITY:
Inclusion Criteria:

* Primary esophageal cancer without known extension beyond the esophagus. (i.e. believed to be Tumor Stage 1-3).
* Scheduled for potentially curative esophageal cancer surgery.
* Written informed consent, including willingness to be randomized to intravenous versus volatile anesthesia.

Exclusion Criteria:

* Previous surgery for esophageal cancer (except diagnostic biopsies) Age <18 or >85 years old.
* ASA Physical Status ≥4.
* Any contraindication to propofol or sevoflurane.
* Other cancer not believed by the attending surgeon to be in long-term remission.
* Systemic disease believed by the attending surgeon to present ≥25% two- year mortality.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1614 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 4 years
  Patients who did not experience cancer recurrence and/or death.

SECONDARY OUTCOMES:
ICU duration | From ICU admission until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 100 months
  Postoperative time in ICU during initial admission.
Hospital duration | Up to 100 months
  Postoperative time spent in hospital during initial admission.
QoR-15 | 2 days
  Quality of Recovery 15 score on postoperative day 2.

CONTACTS AND LOCATIONS:
Overall Officials: Yuwei Oui, MD, Principal Investigator — Shahai Hospital
Locations (1):
- Shanhai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared collaboratively with appropriate approvals and contracts.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 years after publication of the main paper.
Access Criteria: Contact investigators.